CLINICAL TRIAL: NCT02446041
Title: Adherence and COPD Exacerbation Rates in Patients Initiating ICS/LABA Therapy.
Brief Title: ICS/LABA Adherence and COPD Exacerbation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Carelon Research (Other)
Responsible Party: Sponsor
Other Study IDs: D589BR00034
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease; Chronic Obstructive
Keywords: COPD; Chronic Bronchitis; Pulmonary Emphysema
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Pulmonary Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ICS/LABA Patients: ICS/LABA Patients following standard of care
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
The purpose of this retrospective, non-interventional sutdy is to compare the effectiveness of ICS/LABA combination therapy in the reduction of COPD exacerbations during the 12 months after initiation of therapy between COPD patients who are adherent to the index medication and those who are non-adherent.

DETAILED DESCRIPTION:
This retrospective, observational study will assess the effectiveness of ICS/LABA combination therapies among COPD patients new to the ICS/LABA combination therapies in the US, comparing those who are adherent to the index medication and those who are non-adherent. Adherence will be measured using the proportion of days covered with the index medication. Medical and pharmacy claims data will be used as the data source.

ELIGIBILITY:
Inclusion Criteria:

* at least one prescription fill for ICS/LABA combination during identification period.
* COPD diagnosis
* 40 years or older at index date
* > or = 12 months of continuous health plan enrollment prior to and following index date
* 1 or more prescription for SABA, SAMA or SABA/SAMA during the pre-index period.

Exclusion Criteria:

* Patients with prescription claim for ICS/LABA combination therapy during the 12 month pre-index period
* Patients receiving oral corticosteroid medication for more than 180 days during the 12 month pre-index period
* Patients with cancer diagnosis in 12 month pre-index period

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICS/LABA patients with administrative claims data from health plans in the Northeast, Midwest, South and West United States.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate | 12 months
  Rate of COPD exacerbation occurring during the 12 months after therapy initiation.

SECONDARY OUTCOMES:
Severe Exacerbation rate | 12 months
  Severe exacerbation rate during the 12 months after therapy initiation

OTHER OUTCOMES:
Time to Exacerbation | 12 months
  Time to first COPD exacerbation during the 12 months after therapy initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Trudo, MD, Study Chair — AstraZeneca
Locations (1):
- Research Facility, Wilmington, Delaware, United States

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3847&filename=CSR_synopsis.pdf